CLINICAL TRIAL: NCT06398873
Title: Effect of Dupilumab on Nasal Epithelial Barrier Function in Patients With Chronic Rhinosinusitis With Nasal Polyps (CRSwNP) - an Exploratory Pilot Study
Brief Title: Effect of Dupilumab on Nasal Epithelial Barrier Function in Patients With CRSwNP
Acronym: EpiBar
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Sven Schneider, MD, MD, Medical University of Vienna
Other Study IDs: EpiBar
Record Dates: First submitted 2024-04-25; First posted 2024-05-03 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2024-06

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Chronic Rhinosinusitis Without Nasal Polyps
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, primary nasal epithelial cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CRSsNP
- CRSwNP: Dupilumab
  Interventions: Drug: Dupilumab 300 MG/2 ML Subcutaneous Solution [DUPIXENT]

INTERVENTIONS:
Drug: Dupilumab 300 MG/2 ML Subcutaneous Solution [DUPIXENT] — 300mg/2 weeks
  Groups: CRSwNP

SUMMARY:
The investigators aim to investigate two major so far unresolved topics in CRSwNP research: (1) Thorough functional and molecular characterisation of barrier function in patients suffering from CRSsNP and CRSwNP and (2) effect of dupilumab treatment on barrier function in polyp patients. This will be achieved in patient-derived samples by employing measurement of barrier function in primary cell cultures in combination with a mass cytometry based imaging approach, transcriptomic analysis as well as cytokine and microbiome data of individual patients.

DETAILED DESCRIPTION:
Primary objective 1: Characterization of differences in barrier function of the nasal epithelium in patients suffering from CRSsNP, CRSwNP with and without asthma or N-ERD (in absence of therapy with monoclonal antibodies). T Primary objective 2: Effect of dupilumab treatment on barrier function of the nasal epithelium in patients suffering from CRSwNP with and without asthma or N-ERD.

ELIGIBILITY:
Inclusion Criteria:

* 18-99 years of age
* Willingness to participate in the study
* Suffer from chronic rhinosinusitis defined as in EPOS 2020 criteria, see main text
* Group 1 (n=20, CRSsNP): Absence of nasal polyps
* Group 2 (N=60, CRSwNP): Presence of nasal polyps as confirmed by endoscopy or CT and planned therapy with dupilumab
* Presence or absence of non-steroidal anti-inflammatory drug (NSAID)-Exacerbated Respiratory Disease (N-ERD)
* Patients with a history of treatment with monoclonal antibodies will only be included if at least a washout period of 6 months has passed

Exclusion Criteria:

* Pregnancy (as determined by ß-HCG test) or breast feeding
* Patients with severe anatomic variations or deviations that do not allow access to all areas in the nasal cavity
* Patients with cystic fibrosis or primary ciliary dyskinesia
* Patients with permanent immunosuppression
* A mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Patients with clinically meaningful comorbidity as determined by the evaluating committee
* Patients with a history of exacerbation of chronic rhinosinusitis 4 weeks prior to the screening visit
* Intake of a burst of systemic corticosteroids for the treatment of CRS 4 weeks prior to the screening visit

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic rhinosinusitis with and without nasal polyps
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Barrier function in CRSsNP and CRSwNP | 1 Visit (baseline)
  Cell index (xCELLigence)
Barrier function in CRSwNP with Dupilumab | 3 Visits (baseline, 3 months, 6 months)
  Cell index (xCELLigence)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria, Austria

IPD SHARING:
Plan to Share IPD: No
IPD will be shared upon reasonable request

REFERENCES:
- [Background] Bachert C, Han JK, Desrosiers M, Hellings PW, Amin N, Lee SE, Mullol J, Greos LS, Bosso JV, Laidlaw TM, Cervin AU, Maspero JF, Hopkins C, Olze H, Canonica GW, Paggiaro P, Cho SH, Fokkens WJ, Fujieda S, Zhang M, Lu X, Fan C, Draikiwicz S, Kamat SA, Khan A, Pirozzi G, Patel N, Graham NMH, Ruddy M, Staudinger H, Weinreich D, Stahl N, Yancopoulos GD, Mannent LP. Efficacy and safety of dupilumab in patients with severe chronic rhinosinusitis with nasal polyps (LIBERTY NP SINUS-24 and LIBERTY NP SINUS-52): results from two multicentre, randomised, double-blind, placebo-controlled, parallel-group phase 3 trials. Lancet. 2019 Nov 2;394(10209):1638-1650. doi: 10.1016/S0140-6736(19)31881-1. Epub 2019 Sep 19. PMID 31543428
- [Background] Schneider S, Poglitsch K, Morgenstern C, Quint T, Gangl K, Sinz C, Bartosik T, Campion NJ, Liu DT, Landegger LD, Tu A, Stanek V, Rocha-Hasler M, Bangert C, Eckl-Dorna J. Dupilumab increases aspirin tolerance in NSAID-exacerbated respiratory disease. Eur Respir J. 2023 Mar 16;61(3):2201335. doi: 10.1183/13993003.01335-2022. Print 2023 Mar. PMID 36549708